CLINICAL TRIAL: NCT04285931
Title: Prevelance of Dental Caries in Agroup of Egyption Children Using Caries Assessment Spectrum and Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Sabry, demosrator, Cairo University
Other Study IDs: Caries index
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the prevalence of dental caries in Egyptian children aged from 6 to 9 years oldusing CAST index and DMFT index

DETAILED DESCRIPTION:
To explore the prevalence of dental caries in Egyptian children aged from 6 to 9 years oldusing CAST index and DMFT index. from MUST university outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* - Parental or guardian acceptance for participation in the study.
* Children who are medically free from any systemic diseases.
* Children with mixed dentition aging from 6-9 years old.
* Both genders.

Exclusion Criteria:

* uncooperative patient

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be selected from the Outpatients' clinic of Pediatric Dentistr Department, Faculty of Dentistry, Misr University for Science and Technology
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Prevelance of caries using dmft index | 3month
  MDFT index

SECONDARY OUTCOMES:
Prevelance of caries index using cast index | 3 month
  CAST index